CLINICAL TRIAL: NCT06254053
Title: Clinical and Radiographic Evaluation of Zirconomer Restorative Material Versus a Glass Ionomer Cement in Restoration of Primary Molars A Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Zirconomer Restorative
Acronym: Zirconomer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Tamador Ahmed Ibrahim, DR tamador ahmed, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Evaluation of zirconomer; cairo university (Other Grant/Funding Number: faculty of pedatric dentistry)
Record Dates: First submitted 2024-01-30; First posted 2024-02-12 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Dental Caries in Children; Dental Materials
Keywords: GIc/Zirconomer
MeSH Terms: interventions — Glass Ionomer Cements

STUDY DESIGN:
Intervention Model Description: last decade has seen several innovative additions to enhance the properties of GIC whilst simplifying its usage. Unlike the early glass-ionomers, these newer systems are easy and more practical to use as a dental restorative and luting material for preschoolers, children and teenagers alike. These new varieties are composed of ceramic and zirconia reinforced glass ionomer cements were introduced to provide better drawbacks of amalgam as well as tooth-colored restorative materials exhibiting the strength of amalgam and at the same time maintain the fluoride releasing capacity of GIC providing better mechanical properties.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconomer Restorative material in primary molar (Experimental): Arm one zirconomer restorative material (intervention)
  Interventions: Other: zirconia reinforced glass ionomer
- Glass Ionomer Cement in primary molar (Active Comparator): Arm two Glass Ionomer cement (control)
  Interventions: Other: Glass ionomer cement

INTERVENTIONS:
Other: zirconia reinforced glass ionomer — Restorative material
  Other Names: zirconomer
  Arms: Zirconomer Restorative material in primary molar
Other: Glass ionomer cement — Restorative material
  Other Names: GIC
  Arms: Glass Ionomer Cement in primary molar

SUMMARY:
Is zirconomer restorative material more effective than a glass ionomer cement in restoration of primary molars

DETAILED DESCRIPTION:
This trial seeks to evaluate the clinical and radiographic performance of two materials zirconomer restorative material and glass ionomer cement to achieve better treatment for primary molars.

ELIGIBILITY:
* Inclusion criteria:

  1. Children having carious primary molars(class1) without pulp exposure and normal radiograph.
  2. Children between age 5 and 7 years.
  3. Both male and female are included.
  4. Cooperative Children.

     Exclusion criteria:

  <!-- -->

  1. Patients with systemic diseases.
  2. Parent refuse to participate.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-03 (Estimated)

PRIMARY OUTCOMES:
Recurrent CariesColor match | 12 MONTHS
  Radiographic Visual inspection using Modified United States Public Health Service Ryge criteria USPHS

SECONDARY OUTCOMES:
Color match | 12 MONTHS
  visual inspection using Modified United States Public Health Service Ryge criteria USPHS
Marginal Discoloration | 12 MONTHS
  using visual inspection Modified United States Public Health Service Ryge criteria USPHS
Marginal Adaptation | 12 MONTHS
  using visual inspection Modified United States Public Health Service Ryge criteria USPHS
-Anatomic Form | 12 MONTHS
  using visual inspection Modified United States Public Health Service Ryge criteria USPHS

CONTACTS AND LOCATIONS:
Overall Officials: sherien ez zaldein, professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
study protocol and statistical analysis
Supporting Information: Study Protocol, SAP
Time Frame: after one year
Access Criteria: with other investigator including who will work with systematic review ,will provide the clinical study report with the documents above
URL: https://pubmed.ncbi.nlm.nih.gov/34904122/

REFERENCES:
- [Background] Nanavati K, Katge F, Chimata VK, Pradhan D, Kamble A, Patil D. Comparative Evaluation of Shear Bond Strength of Bioactive Restorative Material, Zirconia Reinforced Glass Ionomer Cement and Conventional Glass Ionomer Cement to the Dentinal Surface of Primary Molars: an in vitro Study. J Dent (Shiraz). 2021 Dec;22(4):260-266. doi: 10.30476/DENTJODS.2021.87115.1230. PMID 34904122
- [Background] Kukreja R, Singla S, Bhadoria N, Pawar P, Gupta K, Khandelwal D, Dewani N. An In Vitro Study to Compare the Release of Fluoride from Glass Ionomer Cement (Fuji IX) and Zirconomer. Int J Clin Pediatr Dent. 2022 Jan-Feb;15(1):35-37. doi: 10.5005/jp-journals-10005-2141. PMID 35528493
- [Background] undefined
- [Background] Mushtaq U, Mushtaq F, Thakur D, Rathee K, Poonia N, Khullar S. Comparative Evaluation of Postoperative Sensitivity Following Restoration of Class I Lesions with Different Restorative Materials: An In Vivo Study. J Contemp Dent Pract. 2021 Jun 1;22(6):650-654. PMID 34393122
- [Background] Arora D, Jain M, Suma Sogi HP, Shahi P, Gupta I, Sandhu M. In vivo evaluation of clinical performance of Cention N and glass ionomer cement in proximal restorations of primary molars. J Indian Soc Pedod Prev Dent. 2022 Jan-Mar;40(1):23-29. doi: 10.4103/jisppd.jisppd_108_21. PMID 35439879
- [Background] Albeshti R, Shahid S. Evaluation of Microleakage in Zirconomer(R): A Zirconia Reinforced Glass Ionomer Cement. Acta Stomatol Croat. 2018 Jun;52(2):97-104. doi: 10.15644/asc52/2/2. PMID 30034008